CLINICAL TRIAL: NCT06524726
Title: The International PNH Interest Group PNH Registry
Status: Recruiting | Type: Observational
Sponsor: International PNH Interest Group (Other)
Responsible Party: Sponsor
Other Study IDs: 5674-0001
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PNH; Registry; Patient Registry; Paroxysmal Nocturnal Hemoglobinuria; Anemia, Hemolytic; Anemia; Hematologic Diseases; Myelodysplastic Syndromes; Bone Marrow Diseases; Hemoglobinuria; Hemoglobinuria, Paroxysmal
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Anemia, Hemolytic; Anemia; Hematologic Diseases; Myelodysplastic Syndromes; Bone Marrow Diseases; Hemoglobinuria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PNH patients not receiving anti-complement treatment: PNH patients of any age who are not receiving any anti-complement treatment
- PNH patients receiving anti-complement treatment: PNH patients of any age who are receiving an approved anti-complement treatment

SUMMARY:
The aim of this International PNH Interest Group (IPIG) registry is to develop an international database to prospectively collect data on patients with PNH covering clinical outcomes, patient reported outcomes (PROs), and health-resource utilization (HRU) on all enrolled patients, as well as long term safety data.

DETAILED DESCRIPTION:
The International PNH Interest Group (IPIG) PNH Registry is an international, observational database collecting real-world health information about PNH patients over time. The registry is owned and managed by IPIG, a not-for-profit network of international PNH experts dedicated to improving care and treatment for PNH patients. Several pharmaceutical partners are collaborating with IPIG to fund the registry, which will provide data to support their post-approval regulatory commitments.

The IPIG PNH Registry aims to collect data about all PNH patients including clinical outcomes, patient reported outcomes and health resource usage, as well as long term safety data for patients treated with anti-complement therapies.

The IPIG PNH Registry is comprised of a 'core' PNH disease registry collecting a defined set of core variables on all patients with PNH. In addition, there are several product-specific 'silos' initiated by marketing authorization holders including patients treated with PNH-specific therapies. The silos collect both the core dataset and additional variables to address specific objectives or requests from regulatory authorities (e.g. post-authorization safety data).

Data is collected at enrollment and at 6 monthly intervals during follow-up.

This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44).

ELIGIBILITY:
Inclusion Criteria:

* Patients with PNH confirmed by flow cytometry.
* Patient and/or parent/legally authorized representative provide written informed consent/assent to participate in the registry in a manner approved by the Institutional Review Board/Independent Ethics Committee and local regulations.

Exclusion Criteria:

* Participating in an interventional PNH clinical trial. Note: A patient included in the registry, who enrolls in an interventional PNH clinical trial during the course of the registry, will be kept in the registry but data collection will be paused in the registry during their involvement in the clinical trial/extension study. Data collection in the registry will continue after patient involvement in the clinical trial/extension study has ended or trial protocol mandated data collection ceases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PNH patients with a confirmed diagnosis of PNH by flow cytometry
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2029-05-10 (Estimated); Study Completion 2029-05-10 (Estimated)

PRIMARY OUTCOMES:
Increase knowledge of PNH and describe the PNH patient population | 5-10 years
  To describe PNH disease natural history and PNH treatment course, the patterns of treatment usage, long-term safety of PNH treatments, assess patient reported quality of life and describe health resource usage

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kelly, MBChB PhD, Principal Investigator — International PNH Interest Group; Jeff Szer, MB BS FRACP, Study Chair — International PNH Interest Group
Locations (1):
- International PNH Interest Group, Altamonte Springs, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate information about the registry data will be made available to funding pharmaceutical partners and participating sites in the form of an annual report.

REFERENCES:
- See also: IPIG Website — https://www.pnhinterestgroup.org/